CLINICAL TRIAL: NCT05820399
Title: Ability of Organic Guayusa Extract to Augment Desire to Train, Training Load, and Cardiometabolic Function in Physically Active Women Performing A High Intensity Exercise Training Program
Brief Title: Guayusa Extract on Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathaniel Jenkins (Other)
Responsible Party: Sponsor-Investigator, Nathaniel Jenkins, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 202110443
Record Dates: First submitted 2023-03-24; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Desire to Exercise; Exercise Training; Physical Exertion

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo Controlled, Parallel Arm Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organic Guayusa Extract + High Intensity Exercise (Experimental): Participants will consume an organic guayusa extract supplement that contains caffeine and antioxidants each day for 6 weeks while completing the exercise training program on 3 days/week. On days that participants exercise, they will consume the supplement 30-60 minutes before exercise training. On days they do not exercise, they will consume the capsules upon waking.
  Interventions: Dietary Supplement: Organic Guayusa Extract
- Placebo + High Intensity Exercise (Placebo Comparator): Participants will consume a placebo consisting of maltodextrin each day for 6 weeks while completing the exercise training program. The placebo will be provided in capsule identical in appearance to the active supplement. On days that participants exercise, they will consume the placebo 30-60 minutes before exercise training. On days they do not exercise, they will consume the capsules upon waking.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Organic Guayusa Extract — Supplementation: Participants will supplement daily with organic guayusa extract, which is a caffeinated Amazonian 'super-leaf' belonging to the holly species that contains a very unique blend of polyphenol antioxidants and caffeine (~20% caffeine, 30% chlorogenic acids, 5% catechins) during 6 weeks of high intensity exercise training. Investigators and participants will be blinded to condition.
  Arms: Organic Guayusa Extract + High Intensity Exercise
Dietary Supplement: Placebo — Participants will supplement daily with placebo (maltodextrin). Investigators and participants will be blinded to condition.
  Arms: Placebo + High Intensity Exercise

SUMMARY:
Guayusa extract is a caffeinated Amazonian 'super-leaf' belonging to the holly species that contains a very unique blend of polyphenol antioxidants and caffeine (~20% caffeine, 30% chlorogenic acids, 5% catechins). It is also remarkably low in tannins which are responsible for the bitter taste found in most teas - giving it a sweet flavor profile. As such, it is marketed as an ingredient that can help support energy and performance with potential health-related benefits due to its antioxidant properties. Indeed, ingredients such as these are often consumed by individuals prior to exercise in order to help improve exercise performance, or otherwise to support health-related goals. Whereas several studies have suggested that caffeine and chlorogenic acid consumption may improve performance, mood, and concentration, and some evidence in animals have linked catechin consumption to improved health outcomes, no studies have previous studied whether guayusa extract supplementation helps to support exercise performance in humans. In this study, we will test the whether dietary supplementation with the botanical organic guayusa extract helps support (1) the desire to exercise and exercise performance throughout a 6-week high intensity exercise training program, and thus (2) helps support the physiological adaptations (including body composition, fasting metabolic biomarkers, blood pressure and heart rate, submaximal and maximal exercise performance and fuel metabolism, and changes in the gut microbiome/mycobiome) to a 6-week high intensity exercise training program.

Question 1: Does organic guayusa extract supplementation support the desire to train and training load in physically-active women performing a high-intensity exercise training program?

Question 2: Does organic guayusa extract supplementation support physiological adaptation to exercise (including body composition, fasting metabolic biomarkers, blood pressure and heart rate, submaximal and maximal exercise performance and fuel metabolism, and changes in the gut microbiome/mycobiome) in physically-active women performing a high-intensity exercise training program?

ELIGIBILITY:
Inclusion Criteria:

* Females
* 18-45 years, inclusive
* Physically active >=150 min/wk Moderate Intensity or >=75 min/wk Vigorous Intensity PA) for >=3 months
* BMI < 35 kg/m2
* Otherwise healthy and ready to participate in an exercise program as indicated by responses on the 2021 Physical Activity Readiness Questionnaire Plus (PAR-Q+)
* Habitual caffeine consumption <=200 mg/day OR 2-week washout of current caffeine usage prior to participation
* No current dietary supplementation OR 2-week washout of current supplement usage prior to participation

Exclusion Criteria:

* Current injury or illness that precludes exercise participation
* Current nicotine or cannabis use
* Use of prescription ADD/ADHD, anti-depressant, or other central acting medication, or previously diagnosed ADD/ADHD, clinically depressed, or generalized anxiety disorder
* Current taking prescription stimulants (i.e., Adderall, Ritalin, Vyvanse, etc.)
* Participants with a history of metabolic, hepatorenal, musculoskeletal, autoimmune, or neurologic disease; or currently taking thyroid, hormonal, hyperlipidemic, hypoglycemic, anti-hypertensive, anti-inflammatory, or anti-coagulant medications.
* Treated for Metabolic Syndrome or having been clinically diagnosed with, or taking medication for a cardiometabolic-disorder (e.g., Pre-diabetes, Type II diabetes, high blood pressure, obesity, hypercholesterolemia, etc.)
* Currently pregnant or lactating
* Diagnosed allergy to any ingredient present within the study treatments
* Current competitive NCAA athlete
* Inability or unwillingness to comply with the controls and conditions of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Desire to Exercise | Throughout 6-week training period.
  Desire to Exercise will be assessed Primarily via the Assessment of Exercise Readiness using a 41-item Exercise Readiness Questionnaire.
Exercise Adherence | Throughout 6-week training period.
  Exercise training session adherence will be assessed across all exercise training sessions as a primary quantitative indicator of desire to exercise. Adherence will be assessed as the actual number of completed exercise sessions among participants in each group relative (i.e., percent, %) to the number of total planned exercise sessions. Group differences in session adherence will be compared by chi squared tests.
Exercise Training Load | Throughout 6-week training period.
  Resistance Exercise Training Volume (normalized to bodyweight) will be quantified in each resistance training workout (2x/week) and used as a quantitative indicator of exercise performance/effort.

SECONDARY OUTCOMES:
Desire to Exercise Secondary Measures | Throughout 6-week training period.
  Secondary assessments of Desire to Exercise will include visual analog scales (range 0 - 50, with 0 indicating lower desire and 50 indicating higher desire) used to assess readiness immediately before exercise sessions to "exercise right now", to "invest physical energy right now" and to "invest mental energy right now".
Exercise Training Performance | Throughout 6-week training period.
  Secondary assessments of exercise training performance will include performance during a) a weekly airbike interval exercise session (Avg W), b) a weekly 500 m row (time to completion, Avg W), and c) the time (min) taken to complete the weekly metabolic conditioning workout.
VO2peak | baseline, <7 days after completing the intervention
  VO2peak will be assessed during a ramp test on a electronically-braked cycle ergometer performed to volitional exhaustion with pulmonary gas exchange analysis.
Submaximal Exercise Fat Oxidation | baseline, <7 days after completing the intervention
  Submaximal Exercise Fat Oxidation (%) will be assessed during exercise at a fixed power (i.e., 75W) on an electronically-braked cycle ergometer with pulmonary gas exchange analysis.
Submaximal Exercise Blood Pressure | baseline, <7 days after completing the intervention
  Submaximal Systolic and Diastolic Exercise Blood Pressure (mmHg) will be assessed during exercise at a fixed power (75W) on an electronically-braked cycle ergometer.
Fasting metabolic biomarkers | baseline, <7 days after completing the intervention
  Total cholesterol, HDL-cholesterol, LDL-cholesterol, non-HDL cholesterol, triglycerides, glucose, insulin, c-peptide, GLP-1, GIP
Fasting total cholesterol | baseline, <7 days after completing the intervention
  Total cholesterol will be assessed from a fasting blood sample.
Fasting HDL-cholesterol | baseline, <7 days after completing the intervention
  HDL-cholesterol will be assessed from a fasting blood sample.
Fasting non-HDL cholesterol | baseline, <7 days after completing the intervention
  Non-HDL cholesterol will be assessed from a fasting blood sample.
Fasting triglycerides | baseline, <7 days after completing the intervention
  Triglycerides will be assessed from a fasting blood sample
Fasting Glucose | baseline, <7 days after completing the intervention
  Glucose will be assessed from a fasting blood sample
Fasting insulin | baseline, <7 days after completing the intervention
  insulin will be assessed from a fasting blood sample
Fasting c-peptide | baseline, <7 days after completing the intervention
  Fasting c-peptide will be assessed from a fasting blood sample
Fasting GLP-1 | baseline, <7 days after completing the intervention
  Fasting GLP-1 will be assessed from a fasting blood sample
Fasting GIP | baseline, <7 days after completing the intervention
  Fasting GIP will be assessed from a fasting blood sample
Fasting IL-6 | baseline, at 1 week during the intervention, <7 days after completing the intervention
  IL-6 will be assessed from a fasting blood sample
Fasting IL-10 | baseline, at 1 week during the intervention, <7 days after completing the intervention
  IL-10 will be assessed from a fasting blood sample
Fasting TNFa | baseline, at 1 week during the intervention, <7 days after completing the intervention
  TNFa will be assessed from a fasting blood sample
Fasting triiodothyronine (T3) | baseline, at 1 week during the intervention, <7 days after completing the intervention
  Triiodothyronine (T3) will be assessed from a fasting blood sample
Fasting thyroxine (T4) | baseline, at 1 week during the intervention, <7 days after completing the intervention
  Thyroxine (T4) will be assessed from a fasting blood sample
Fasting Progesterone | baseline, at 1 week during the intervention, <7 days after completing the intervention
  Progesterone will be assessed from a fasting blood sample
Fasting Testosterone | baseline, at 1 week during the intervention, <7 days after completing the intervention
  Testosterone will be assessed from a fasting blood sample
Fasting Estrogen | baseline, at 1 week during the intervention, <7 days after completing the intervention
  Estrogen will be assessed from a fasting blood sample
Fasting Cortisol | baseline, at 1 week during the intervention, <7 days after completing the intervention
  Cortisol will be assessed from a fasting blood sample
Fasting Adiponectin | baseline, <7 days after completing the intervention
  Adiponectin will be assessed from a fasting blood sample
Fasting Leptin | baseline, <7 days after completing the intervention
  Leptin will be assessed from a fasting blood sample
Fasting Adipsin | baseline, <7 days after completing the intervention
  Adipsin will be assessed from a fasting blood sample
Fasting Lipocalin | baseline, <7 days after completing the intervention
  Lipocalin will be assessed from a fasting blood sample
Fasting Plasminogen activator inhibitor-1 (PAI-1) | baseline, <7 days after completing the intervention
  Plasminogen activator inhibitor-1 (PAI-1) will be assessed from a fasting blood sample
Fasting Resistin | baseline, <7 days after completing the intervention
  Resistin will be assessed from a fasting blood sample

OTHER OUTCOMES:
Rating of Perceived Exertion | Throughout 6-week training period.
  RPE will be assessed following each exercise session to determine subjective effort for each session on a scale of 1-10, where 1 is lowest perceived effort (e.g., rest) and 10 is greatest perceived effort.

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Laboratory of Applied Physiology and Lifestyle Medicine, Iowa City, Iowa, United States